CLINICAL TRIAL: NCT06112717
Title: The Application of the Self Care Deficit Nursing Theory in Adolescents With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tuğçe TORUN, PhD, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HACETTEPEU-TUGCETORUN-001
Record Dates: First submitted 2023-10-29; First posted 2023-11-01 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis; Adolescence; Self-care
Keywords: Cystic Fibrosis; Adolescence; Self-care
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: There are 2 group in the study. Intervention Group and Control Group. The control group received no intervention by principal researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing Care (Experimental): Seven home visit was made to adolescent in the intervention group. In the first and last visits only self-care knowledge and skills of adolescents were evaluated. In the 2.,3.,4.,5. and 6. home visits they received supportive-educational individualised nursing care based on Orem's Self Care Deficit Nursing Theory. The applied nursing interventions varied based on the individual needs and the level of assistance required by each adolescent. Each home visit lasted 30-60 minutes. Adolescents were given an educational booklet containing information about self-care in cystic fibrosis.
  Interventions: Other: Supportive-Educative Nursing Care
- Control Group (No Intervention): Adolescents in the control group received no intervention by the researcher.

INTERVENTIONS:
Other: Supportive-Educative Nursing Care — Adolescents in the intervention group were received Supportive-Educative Nursing Care based on Orem's Self Care Deficit Nursing Theory
  Arms: Nursing Care

SUMMARY:
The present study evaluates the effect of nursing care based on the Self-Care Deficit Nursing Theory on the knowledge and skills related to self-care among adolescents with Cystic Fibrosis.

DETAILED DESCRIPTION:
This study included 30 adolescents who were equally divided into the intervention and control groups. The data were collected by using the Sociodemographic Data Form and the Self-Care Knowledge and Skills Evaluation Forms for Adolescents with Cystic Fibrosis. A total of seven home visits were conducted with the adolescents in the intervention group, during which individualized care plans were applied based on the Self-Care Deficit Nursing Theory. The self-care needs of the adolescents in the control group were identified based on data collected during two home visits conducted at the onset of the study and after 4.5 months.

As a result of the application of nursing interventions based on the Self-Care Deficit Nursing Theory, a statistically significant increase was noted in the self-care knowledge and skills of the adolescents in the intervention group (p<0.05). Additionally, nursing interventions and nursing diagnosis decreased significantly over time in all adolescents in the intervention group (p<0.05).

Orem's Self-Care Deficit Nursing Theory was useful in enhancing the self-care knowledge and skills of adolescents with Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis determined by a positive sweat test and/or the presence of two Cystic Fibrosis mutations,
* Aged between 12 and 18 years
* Living in the same Ankara

Exclusion Criteria:

* Adolescents with mental health issues
* Adolescents with an atypical form of Cystic Fibrosis (characterized by an absence of symptoms and no medication requirement)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The change in self care knowledge and skills of adolescents with Cystic Fibrosis | 18 weeks(4.5 months) after first enrollment of patient.
  The change in self-care knowledge and skills of adolescents at the end of the research after the applied nursing interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Çavuşoğlu, Professor, Study Director — Head of Pediatric Nursing Department, Faculty of Nursing, Hacettepe University, Turkey; Deniz Doğru, Professor, Study Director — Pediatric Pulmonology Department, Faculty of Medicine, Hacettepe University, Turkey; Tuğçe TORUN, PhD, Principal Investigator — Pediatric Nursing Department, Faculty of Nursing, Hacettepe University, Turkey
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No